CLINICAL TRIAL: NCT04383847
Title: Understanding the Role of Gender Inequality and Food Insecurity on Maternal and Child Health
Acronym: K01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Center for Research on Environment, Health and Population Activities (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DiamondSmithK01; K01HD086281 (NIH)
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Feasibility study in 30 groups, pre post, no control
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main study (Experimental): There is only 1 arm because this is a feasibility and acceptability pilot.
  Interventions: Behavioral: Sumadhur Aarambha

INTERVENTIONS:
Behavioral: Sumadhur Aarambha — Group intervention for newly married women, their husbands, and mothers-in-law with information mainly about nutrition, but also pre-pregnancy health, reproductive/pregnancy health and gender equality.

SUMMARY:
To pilot test a group intervention for newly married women and their households to improve nutrition, pregnancy and delivery knowledge, and intrahousehold communication

DETAILED DESCRIPTION:
Aim: To test the feasibility of an empowerment and food insecurity intervention for newly married women and others in their households to improve maternal and child health outcomes. The investigators will pilot an intervention consisting of groups of newly married women, their husbands and mothers-in-law. Each household will be enrolled for 4 months in weekly sessions. Topics discussed will include behavioral messaging crafted specifically for newly married households (including husbands and in-laws) to address the perceptions of different family members about food consumption, gender inequality, and the relationship between women's nutrition, food consumption, maternal health, and birth outcomes. Behavioral messaging at the household level: Based on findings from preliminary studies, key barriers to newly married women receiving needed nutrition/food and potential mechanisms to address those barriers were identified, as well as informational messages that could be used to address specific barriers. Particular attention was paid to how household dynamics and decision-making relate to gender inequality and food insecurity. Thirty randomly selected newly married households will be recruited to participate in testing the feasibility and acceptability of the intervention. Acceptability will be assessed from women, husbands, and mothers-in-law through surveys at the end of 4 months with questions on relevance to their needs, information gained, and interest in participating further. Enrollment and retention at 4 months will also be used to measure acceptability. Preliminary changes in knowledge, attitudes and behaviors will be assessed through a comparison of pre and post survey data. The investigators will also conduct semi structured interviews with 15 participants and 5 stakeholders. If necessary, the intervention will then be refined.

ELIGIBILITY:
Inclusion Criteria:

* the household has a newly married couple (married in the last 3 months)
* a living mother-in-law
* both the woman and man being over the age of 18

Exclusion Criteria:

* Under 18
* not recently married

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Attendance and Attrition of Participants | 4 months
  Proportion of meetings that respondents reported that they attend, combined with the attrition rate
Participant Satisfaction | 4 months
  Proportion of respondents who state that they were satisfied with the intervention, answering "Very satisfied" or "satisfied" to a 5 point scale from very dissatisfied, dissatisfied, neither dissatisfied or satisfied, satisfied or very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia G Diamond-Smith, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community based, Nawalparasi, Nawalparasi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diamond-Smith N, Mitchell A, Cornell A, Dahal M, Gopalakrishnan L, Johnson M, Weiser S, Puri M. The development and feasibility of a group-based household-level intervention to improve preconception nutrition in Nawalparasi district of Nepal. BMC Public Health. 2022 Apr 6;22(1):666. doi: 10.1186/s12889-022-12980-w. PMID 35387647